CLINICAL TRIAL: NCT07127016
Title: Mindfulness in Nonflaccid Facial Paralysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00126997
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-07

CONDITIONS: Facial Paralysis
Keywords: non-flaccid facial paralysis; synkinesis; mindfulness
MeSH Terms: conditions — Facial Paralysis; Synkinesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Sessions (Experimental): 8 sessions of mindfulness prior to completing their physical therapy session
  Interventions: Behavioral: Mindfulness Sessions
- No Mindfulness Sessions (Active Comparator): Standard of care no mindfulness sessions
  Interventions: Behavioral: No Mindfulness Sessions

INTERVENTIONS:
Behavioral: Mindfulness Sessions — 8 sessions of mindfulness prior to completing their physical therapy session. Each mindfulness session will take 5-10 minutes and will be completed once weekly, immediately prior to their physical therapy sessions. Mindfulness prompts will focus on self-reflection, relaxation, body scanning and being present.
  Arms: Mindfulness Sessions
Behavioral: No Mindfulness Sessions — Standard of care physical therapy without mindfulness sessions.
  Arms: No Mindfulness Sessions

SUMMARY:
The purpose of this study is to learn more about how mindfulness techniques can help reduce anxiety, depression and body image disturbance as well as improve synkinesis in individuals with non-flaccid facial paralysis.

DETAILED DESCRIPTION:
This study will utilize a prospective randomized two-arm intervention design to assess the effects of mindfulness on patients with non-flaccid facial paralysis. Patients will either be randomized to the normal standard of care Physical Therapy intervention for 8 weeks, or Physical therapy and 8 sessions of mindfulness for 8 weeks. The patients randomized to the mindfulness intervention will undergo 8 sessions of mindfulness prior to completing their physical therapy session. These mindfulness interventions will be recordings administered through a phone or computer, through mindfulsynkinesis.com. Mindfulness scripts were created using Open Network materials and verified by a medical doctor and physical therapist trained in Mindfulness Based Stress Reduction. Each mindfulness session will take 5-10 minutes and will be completed once weekly, immediately prior to their physical therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with non-flaccid facial paralysis (NFFP) due to Bell's Palsy, Ramsay Hunt syndrome, Lyme disease, or post-acoustic neuroma resection, at least 8 months from the initial diagnosis

Exclusion Criteria:

* Received treatments such as botox or physical therapy for facial paralysis
* History of malignancy or facial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Facial Clinimetric Evaluation Scale (FaCE) | Baseline
  15 items rated on a 5-point Likert scale where 1 corresponds to the lowest level of function and 5 corresponds to the highest level of function. The items are categorized into 6 domains: facial movement, facial comfort, oral function, eye comfort, lacrimal control and social function with each domain being scored out of a total of 100 where 0 is the worst possible score to 100 being the best. The mean derived from all domains will determine the total score (out of 100).
Facial Clinimetric Evaluation Scale (FaCE) | Week 8
  15 items rated on a 5-point Likert scale where 1 corresponds to the lowest level of function and 5 corresponds to the highest level of function. The items are categorized into 6 domains: facial movement, facial comfort, oral function, eye comfort, lacrimal control and social function with each domain being scored out of a total of 100 where 0 is the worst possible score to 100 being the best. The mean derived from all domains will determine the total score (out of 100).
Facial Clinimetric Evaluation Scale (FaCE) | Week 16
  15 items rated on a 5-point Likert scale where 1 corresponds to the lowest level of function and 5 corresponds to the highest level of function. The items are categorized into 6 domains: facial movement, facial comfort, oral function, eye comfort, lacrimal control and social function with each domain being scored out of a total of 100 where 0 is the worst possible score to 100 being the best. The mean derived from all domains will determine the total score (out of 100).
Hospital Anxiety and Depression Scale (HADS) | Baseline
  14-item questionnaire measuring anxiety and depression levels. Total score range is 0-21 with higher score indicating higher likelihood of anxiety/depression.
Hospital Anxiety and Depression Scale (HADS) | Week 8
  14-item questionnaire measuring anxiety and depression levels. Total score range is 0-21 with higher score indicating higher likelihood of anxiety/depression.
Hospital Anxiety and Depression Scale (HADS) | Week 16
  14-item questionnaire measuring anxiety and depression levels. Total score range is 0-21 with higher score indicating higher likelihood of anxiety/depression.
Synkinesis Assessment Questionnaire (SAQ) | Baseline
  9-item questionnaire assessing patient perceived severity of synkinesis using a five-point scale. Total score ranges from 20-100. High score means a greater perceived severity of synkinesis symptoms, low score means less perceived severity of synkinesis symptoms.
Synkinesis Assessment Questionnaire (SAQ) | Week 8
  9-item questionnaire assessing patient perceived severity of synkinesis using a five-point scale. Total score ranges from 20-100. High score means a greater perceived severity of synkinesis symptoms, low score means less perceived severity of synkinesis symptoms.
Synkinesis Assessment Questionnaire (SAQ) | Week 16
  9-item questionnaire assessing patient perceived severity of synkinesis using a five-point scale. Total score ranges from 20-100. High score means a greater perceived severity of synkinesis symptoms, low score means less perceived severity of synkinesis symptoms.
Mindfulness Attention Awareness Scale (MAAS) | Baseline
  15-item questionnaire to assess a core characteristic of mindfulness and how much you experience mindfulness in everyday life, not just during meditation. Total score range is 15-90. High score indicates more mindful, more likely to be aware of your thoughts, feelings, and sensations in the present moment. Low score indicates less mindful, more distracted or on "automatic pilot."
Mindfulness Attention Awareness Scale (MAAS) | Week 8
  15-item questionnaire to assess a core characteristic of mindfulness and how much you experience mindfulness in everyday life, not just during meditation. Total score range is 15-90. High score indicates more mindful, more likely to be aware of your thoughts, feelings, and sensations in the present moment. Low score indicates less mindful, more distracted or on "automatic pilot."
Mindfulness Attention Awareness Scale (MAAS) | Week 16
  15-item questionnaire to assess a core characteristic of mindfulness and how much you experience mindfulness in everyday life, not just during meditation. Total score range is 15-90. High score indicates more mindful, more likely to be aware of your thoughts, feelings, and sensations in the present moment. Low score indicates less mindful, more distracted or on "automatic pilot."

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gossett, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No